CLINICAL TRIAL: NCT02394314
Title: A Phase 1, Single-ascending-dose Study to Evaluate the Safety and Pharmacokinetics of MEDI0382 in Healthy Volunteers
Brief Title: A Phase 1, Single Dose Study to Evaluate the Safety and Pharmacokinetics of MEDI0382 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: D5670C00001
Record Dates: First submitted 2015-02-26; First posted 2015-03-20 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers
Keywords: MEDI0382, diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Drug: Placebo
- MEDI0382 (Experimental): MEDI0382 administered subcutaneously
  Interventions: Drug: MEDI0382

INTERVENTIONS:
Drug: MEDI0382 — MEDI0382 administered subcutaneously
  Arms: MEDI0382
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
A Phase 1, single dose study with 8 cohorts of ascending doses designed to evaluate the safety and pharmacokinetics of MEDI0382 in healthy volunteers.

DETAILED DESCRIPTION:
This is a first-time-in-humans (FTIH), randomized, double-blind study designed to evaluate the safety, tolerability, and PK of MEDI0382 administered as single-ascending SC doses to healthy subjects (age 18-45). Eight subjects per cohort will be enrolled in a total of 8 cohorts. The decision whether or not to dose escalate will be based upon data review by the Dose Escalation Committee (DEC). Within each cohort, the subjects will be randomized to MEDI0382 or placebo (3:1). Following screening, the study duration for each subject will be approximately 29 days, consisting of an inpatient evaluation period, and an outpatient follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers, ages 18-45
* Must provide written informed consent
* BMI >22 and <30 kg/m2 and body weight >70kg
* Venous access suitable for multiple cannulations
* Vital signs within normal specified ranges
* Females must be non-lactating and non-childbearing potential
* Males must practice 2 effective contraceptive measures if sexually active

Exclusion Criteria:

* Any concurrent condition that in the opinion of the investigator would interfere with the evaluation of the investigational product
* History or presence of gastrointestinal, renal, or hepatic disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* History of cancer, with the exception of non-melanoma skin cancer
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks prior to dosing
* Positive Hepatitis B, Hepatitis C or HIV test or use of antiretroviral medications at screening.
* Concurrent or previous use of a GLP-1 receptor agonist
* Current or previous use of systemic corticosteroids within the past 28 days prior to screening
* Use of any medicinal products or herbal preparations licensed for control of body weight or appetite is prohibited.
* Known or suspected history of alcohol or drug abuse within the past 3 years.
* Positive drug screen
* Current smoker

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 362 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability of MEDI0382 | 28 days post dosing
  Treatment emergent adverse events (TEAEs) and serious adverse events (STEAEs)
Number of subjects with Adverse events as a measure of safety and tolerability of MEDI0382 | 28 days post dosing
  GI symptomatology (a composite of nausea and vomiting)
Number of subjects with Adverse events as a measure of safety and tolerability of MEDI0382 | 28 days post dosing
  Vital signs (systolic and diastolic blood pressure, pulse rate, temperature, and respiratory rate)
Number of subjects with Adverse events as a measure of safety and tolerability of MEDI0382 | 28 days post dosing
  12 lead electrocardiogram including RR, PR, QRS, QT and QTc intervals
Number of subjects with Adverse events as a measure of safety and tolerability of MEDI0382 | 28 days post dosing
  Clinical laboratory assessments (serum chemistry, hematology, urinalysis)

SECONDARY OUTCOMES:
Pharmacokinetics of MEDI0382, maximum plasma concentration (Cmax) | 72 hours postdose
  This variable will be estimated for MEDI0382 where the data allow.
Pharmacokinetics of MEDI0382, area under the curve concentration (AUC) | 72 hours post dose
  This variable will be estimated for MEDI0382 where the data allow.
Proportion of subjects with ADA to MEDI0382 | 28 days post dose
  This variable will be estimated for MEDI0382 where the data allow.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany